CLINICAL TRIAL: NCT02704767
Title: Tarceva With or Without Apatinib in the First-line Therapy of Advanced Lung Adenocarcinoma With Mutant EGFR:a Phase II Study.
Brief Title: Tarceva With or Without Apatinib in the Advanced Lung Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Li Rong-qing, Professor, First Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1stKunmingMC; KMMURO001 (Other: 1stKunmingMU)
Record Dates: First submitted 2016-02-27; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — apatinib; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TarceP (Placebo Comparator): Tarceva with Placebo
  Interventions: Drug: Tarceva; Drug: Placebo
- TarceA (Experimental): Tarceva with Apatinib
  Interventions: Drug: Apatinib; Drug: Tarceva

INTERVENTIONS:
Drug: Apatinib — a tyrosine kinase inhibitor of VEGF invented by Hengrui pharma in China
  Other Names: AiTan
  Arms: TarceA
Drug: Tarceva
Drug: Placebo
  Arms: TarceP

SUMMARY:
Tarceva now was established first-line therapy for advanced lung adenocarcinoma with mutant EGFR patients.However,the benefit lasted for about 6-8 months.So we consider to add apatinib,a tyrosine kinase inhibitor of VEGF,to the therapy of these patients.

DETAILED DESCRIPTION:
Lung adenocarcinoma is the most common NSCLC,most patient were diagnosed to advanced stage.The first-line therapy include chemotherapy of targeted therapy .Tarceva now was established first-line therapy for advanced lung adenocarcinoma with mutant EGFR patients.However,the benefit lasted for about 6-8 months.So we consider to add apatinib,a tyrosine kinase inhibitor of VEGF,to the therapy of these patients.We designed the study to find out whether the addition of apatinib to the Tarceva would enhance the efficacy of Tarceva.

ELIGIBILITY:
Inclusion Criteria:

* lung adenocarcinoma proved by histology;with mutant EGFR;ECOG PS 0-2;Clinical stage IIIb or IV;without other fatal disease;without hemorrhagic disease;normal liver,renal and bone marrow function,not pregnant.

Exclusion Criteria:

* ECOG PS 3-5;abnormal liver,renal and bone marrow function,pregnant;with severe diseases;wild type EGFR

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, assessed up to 36 months
  From date of randomization until the date of death from any cause, assessed up to 36 months
Response rate | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Baas P, Belderbos JS, van den Heuvel M. Chemoradiation therapy in nonsmall cell lung cancer. Curr Opin Oncol. 2011 Mar;23(2):140-9. doi: 10.1097/CCO.0b013e328341eed6. PMID 21178617
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Erlotinib versus chemotherapy as first-line treatment for patients with advanced EGFR mutation-positive non-small-cell lung cancer (OPTIMAL, CTONG-0802): a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2011 Aug;12(8):735-42. doi: 10.1016/S1470-2045(11)70184-X. Epub 2011 Jul 23. PMID 21783417
- [Background] Xu JL, Jin B, Ren ZH, Lou YQ, Zhou ZR, Yang QZ, Han BH. Chemotherapy plus Erlotinib versus Chemotherapy Alone for Treating Advanced Non-Small Cell Lung Cancer: A Meta-Analysis. PLoS One. 2015 Jul 6;10(7):e0131278. doi: 10.1371/journal.pone.0131278. eCollection 2015. PMID 26147288
- [Background] Li H, Takayama K, Wang S, Shiraishi Y, Gotanda K, Harada T, Furuyama K, Iwama E, Ieiri I, Okamoto I, Nakanishi Y. Addition of bevacizumab enhances antitumor activity of erlotinib against non-small cell lung cancer xenografts depending on VEGF expression. Cancer Chemother Pharmacol. 2014 Dec;74(6):1297-305. doi: 10.1007/s00280-014-2610-x. Epub 2014 Oct 26. PMID 25344762
- [Background] Seto T, Kato T, Nishio M, Goto K, Atagi S, Hosomi Y, Yamamoto N, Hida T, Maemondo M, Nakagawa K, Nagase S, Okamoto I, Yamanaka T, Tajima K, Harada R, Fukuoka M, Yamamoto N. Erlotinib alone or with bevacizumab as first-line therapy in patients with advanced non-squamous non-small-cell lung cancer harbouring EGFR mutations (JO25567): an open-label, randomised, multicentre, phase 2 study. Lancet Oncol. 2014 Oct;15(11):1236-44. doi: 10.1016/S1470-2045(14)70381-X. Epub 2014 Aug 27. PMID 25175099
- [Background] Spigel DR, Burris HA 3rd, Greco FA, Shipley DL, Friedman EK, Waterhouse DM, Whorf RC, Mitchell RB, Daniel DB, Zangmeister J, Bass JD, Hainsworth JD. Randomized, double-blind, placebo-controlled, phase II trial of sorafenib and erlotinib or erlotinib alone in previously treated advanced non-small-cell lung cancer. J Clin Oncol. 2011 Jun 20;29(18):2582-9. doi: 10.1200/JCO.2010.30.7678. Epub 2011 May 16. PMID 21576636
- [Background] Scagliotti GV, Krzakowski M, Szczesna A, Strausz J, Makhson A, Reck M, Wierzbicki RF, Albert I, Thomas M, Miziara JE, Papai ZS, Karaseva N, Thongprasert S, Portulas ED, von Pawel J, Zhang K, Selaru P, Tye L, Chao RC, Govindan R. Sunitinib plus erlotinib versus placebo plus erlotinib in patients with previously treated advanced non-small-cell lung cancer: a phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2070-8. doi: 10.1200/JCO.2011.39.2993. Epub 2012 May 7. PMID 22564989
- [Background] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952
- [Background] Hu X, Zhang J, Xu B, Jiang Z, Ragaz J, Tong Z, Zhang Q, Wang X, Feng J, Pang D, Fan M, Li J, Wang B, Wang Z, Zhang Q, Sun S, Liao C. Multicenter phase II study of apatinib, a novel VEGFR inhibitor in heavily pretreated patients with metastatic triple-negative breast cancer. Int J Cancer. 2014 Oct 15;135(8):1961-9. doi: 10.1002/ijc.28829. Epub 2014 Mar 20. PMID 24604288
- [Background] Qin S. Phase III study of apatinib in advanced gastric cancer: a randomized, double-blind, placebo-controlled trial. J Clin Oncol. 2014; 32(Suppl):Abst 4003.
- [Background] Zhang L, Shi M, Huang C, et al. A phase II, multicenter, placebo-controlled trial of apatinib in patients with advanced nonsquamous non-small cell lung cancer (NSCLC) after two previous treatment regimens. J Clin Oncol. 2012;30(Suppl):Abst 7548.